CLINICAL TRIAL: NCT05689424
Title: Suppression of Endogenous Glucose Production by Injectable HDV-Insulin Lispro: A Dose Response Study in Human Subjects With Type 1 Diabetes
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Principal Investigator, Jeremy Pettus, MD, Assistant Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: DP 01-2022-02
Record Dates: First submitted 2023-01-09; First posted 2023-01-19 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- HDV-bound Lispro 0% (Placebo Comparator): Subjects will receive insulin lispro with 0% bound HDV
  Interventions: Drug: HDV-Insulin Lispro
- HDV-bound Lispro 1% (Active Comparator): Subjects will receive insulin lispro with 1% bound HDV
  Interventions: Drug: HDV-Insulin Lispro
- HDV-bound Lispro 10% (Active Comparator): Subjects will receive insulin lispro with 10% bound HDV
  Interventions: Drug: HDV-Insulin Lispro
- HDV-bound Lispro 100% (Active Comparator): Subjects will receive insulin lispro with 100% bound HDV
  Interventions: Drug: HDV-Insulin Lispro

INTERVENTIONS:
Drug: HDV-Insulin Lispro — The name of the investigational drug is Hepatic Directed Vesicles + Insulin Lispro (HDV-bound LIS). It is a nano-carrier-based formulation of insulin which is the active therapeutic ingredient in the product. The nano-carrier component of the formulation contains a hepatic target molecule, biotin phosphatidylethanolamine, which has an affinity for hepatocytes and enables the product to deliver insulin directly to the liver.

SUMMARY:
Single-center, double-blind, random-sequence study assessing the HDV dose-response relationship to Endogenous Glucose Production (EGP), Free Fatty Acids (FFA) and Glucose Disposal Rate (GDR) during a euglycemic clamp procedure following overnight stabilization of blood glucose with intravenous insulin (and, if needed intravenous glucose). EGP and GDR will be determined using established radioisotope methodology. The concentration of Hepatic Directed Vesicles (HDV) in the insulin lispro (LIS) infused during the clamp procedure will be varied such that the percentage of HDV-bound LIS will range from 0%, 1%, 10%, and 100%. Each participant will thus undergo four clamp procedures at the four different HDV levels. LIS will be infused at a constant dose (6 mU/m2/min) for each of the four procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of age 18 to 65 years, inclusive, who:
2. Has at Screening been diagnosed as T1D for at least 12 months; preference will be given to potential participants who currently use continuous subcutaneous insulin infusion (CSII) therapy;
3. Has at Screening C-peptide ≤0.8 ng/mL (single retest allowed);
4. Has at Screening a BMI ≥18.0 kg/m2 and ≤33.0 kg/m2;
5. Has at Screening HbA1c ≥6.5% and ≤8.5 %.

Exclusion Criteria:

1. Has known or suspected allergy to any component of any of the study drugs in this trial;
2. Is, at Screening, pregnant or breast-feeding, or intends to become pregnant at any time during the duration of the study;
3. Has, at Screening, as judged by the Site Investigator, a history or current evidence of any of advance complications of diabetes;
4. Is, at Screening, judged by the Site Investigator to have a current addiction to alcohol or substances of abuse;
5. Is, at Screening, using one or more drugs that may interfere with the interpretation of trial results or are known to cause clinically relevant interference with insulin action, glucose utilization, or recovery from hypoglycemia (e.g., beta blockers, systemic corticosteroids at pharmacologic doses, cancer chemotherapies);
6. Has, within one (1) month prior to Screening, used either oral anti-diabetic medication or noninsulin anti-diabetic injection therapies (e.g. SGLT-2 inhibitors, pramlintide, GLP-1 agonists, etc.);
7. Has, within one (1) month prior to Screening, received any investigational drug;
8. Has, within three (3) months prior to Screening, smoked tobacco or used any smokeless tobacco or nicotine delivery system (inhaled, oral or buccal);
9. Has at Screening, as judged by the Site Investigator, any condition (intrinsic or extrinsic) that could reasonably be expected to interfere with trial participation, confound evaluation of the data, or pose additional risk to adhering to the study protocol. Examples of such conditions include but are not limited to:

   * Clinically significant active disease of the gastrointestinal, cardiovascular, hepatic, neurological, renal, genitourinary, or hematological systems;
   * History of such an illness or disease;
   * Diminished mental capacity, psychological or behavioral dysfunction, unwilling or resistant to protocol requirements, language barriers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of suppression of endogenous glucose production | 0 through 6 hours
  To establish the dose-response relationship between Hepatic-Directed Vesicles (HDV) and endogenous glucose production at a constant dose of insulin lispro (LIS) during euglycemic clamp procedure

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared